CLINICAL TRIAL: NCT01610271
Title: Air Barrier System to Reduce Contamination of Wounds During Surgery
Brief Title: Air Barrier System for the Prevention of Surgical Site Infection
Acronym: ABS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nimbic Systems, LLC (Industry)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH); Baylor College of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: H-28131; 2R44GM095005-02A1 (NIH)
Record Dates: First submitted 2012-05-03; First posted 2012-06-04 (Estimated); Results first posted 2018-12-12 (Actual); Last update posted 2019-01-03 (Actual); Status verified 2018-12

CONDITIONS: Surgical Site Infection
Keywords: Prevention; Surgical Site Infection; Air Barrier System; Implant Infection
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Air Barrier System (Experimental): The Air Barrier System will be employed throughout the surgical procedure for this group of patients.
  Interventions: Device: Air Barrier System
- Control (No Intervention): The Air Barrier System will not be used during the surgical procedure for this group of patients.

INTERVENTIONS:
Device: Air Barrier System — ABS is a device that emits a stream of purified air over the surgical site creating a barrier that prevents the intrusion of bacteria.
  Other Names: ABS
  Arms: Air Barrier System

SUMMARY:
Airborne particles are present in all indoor environments including the operating room. Most of these particles come from the surgical staff moving around in the room, positioning of the patient during surgery, and the movement of surgical equipment and supplies. While the amount of particulate in an operating room is much, much less than is found in a typical home or public space, some particulate is usually present no matter how the room and air are cleaned and filtered. Typically these few particulate cause no problems, but the goal is always to have the cleanest air possible during surgery. The Air Barrier System (ABS) consists of a reusable blower and a sterile nozzle. The blower feeds filtered air into the sterile disposable nozzle, which disperses a constant stream of gentle, high purity air over the surgical incision. This stream of air forms a shield over the surgical area to prevent airborne particulate from settling into the open wound. This is particularly critical for long-duration surgeries, such as procedures that involve the implantation of a prosthesis. The main objective of this research study is to determine whether the ABS can reduce the potential for surgical site infection during total hip replacement, spinal fusion, or lower extremity bypass grafting procedures. These procedures were chosen because each is a long-duration procedure which involves implantation of prosthesis.

DETAILED DESCRIPTION:
Surgical site infection (SSI) following prosthesis implantation and other invasive procedures is a serious complication leading to increased mortality, morbidity, and financial cost to patients and the U.S. healthcare infrastructure. Multiple studies have shown that the primary source of surgical site bacterial colonization is staphylococci shed from the skin of people present in the surgical theatre. These bacteria-carrying skin cells are aerosolized into the environment and deposit into surgical incisions.

The innovations currently pursued in research and industry to combat nosocomial infection fall primarily into three categories: (1) developing new antimicrobial drugs and agents, (2) developing antimicrobial coatings for devices, and (3) implementing procedures to reduce the risk of cross-contamination. Significant resources are being allocated to prevent infections from developing post-operatively and to mitigate the effects of infection once microorganisms enter the body. However, there is little development of new technologies that can be employed in the operating room to prevent the initial intrusion into the surgery site.

All modern surgical theatres utilize some form of air filtration. In a conventional flow system, air streams mix freely in the room. In an OR designed for laminar flow (LFOR), air emits from filters and proceeds into the room in relatively coherent streams. The benefit thought to be achieved by a LFOR, in principle, is that filtered air does not mix with contaminated air before reaching the surgery area. The difficulty in achieving the desired results in a LFOR lies in the fact that once the flow pattern enters the room, it is subjected to a very complex set of dynamics over a significant distance. Air is clean upon leaving the filter bank, but it enters a space laden with airborne bacteria and particulate matter shed from people in the OR.

Nimbic Systems has developed a device, the Air Barrier System (ABS), which shields surgical sites from airborne contaminants in the operating room by creating a localized clean air field directly adjacent to and surrounding the incision site. The ABS consists of two components: a Filter and an air Nozzle with attached Hose. The Filter is a nonsterile reusable component which filters ambient operating room air and forces it through an exit port on the top of the unit. The Nozzle is attached on top of the incision drape adjacent to a surgical incision with Velcro® fastening pads. The end of the Hose is plugged into the Filter's air exit port. Contaminant-free air then flows through the Hose and Nozzle over the incision site. The ABS maintains this protective envelope of bacteria-free air over a wide range of patient and incision site geometries, yet the insertion of hands and instruments are not disrupted by the protective envelope.

The ABS technology was extremely successful at reducing the presence of bacteria and other colony forming units at incision sites during Phase I study. In a randomized, prospective clinical study of 36 hip arthroplasty procedures, the ABS reduced the presence of colony forming units at incision sites by 84% versus ambient operating room levels.

This will be a prospective randomized double-blind pilot trial of the ABS in three surgical specialty applications (total hip arthroplasty, lumbar laminectomy with instrumentation, and femoral-popliteal bypass graft). A cohort of 300 recruited patients will be randomly assigned, at a 1:1 ratio, to either a control group (no ABS) or experimental group (with ABS). The primary outcome of the trial is the occurrence of SSI by one year after surgery using the established CDC definitions and classifications of surgical site infection. Secondary outcomes include (1) measuring levels of colony forming units (CFU) present in the operating room air during surgical procedures to examine correlations with occurrence of SSI; (2) examining types of organisms that cause SSI in the two study groups; and (3) surgeon satisfaction with the ABS device. Patient characteristics and measures of operating room environment will be collected during surgery, and the patients' surgical sites will be clinically evaluated following surgery to identify potential superficial or deep SSI up to one year after surgery. The estimated occurrence of SSI in the control group is 6%, based on baseline data pertaining to the three studied types of surgery at the Michael E. DeBakey VA Medical Center. The anticipated rate of SSI in the experimental group is 3%. The proposed pilot study is designed to detect a clinically relevant reduction (i.e., a 50% reduction, from 6% to 3%) in the observed rate of SSI in patients who are exposed to the ABS vs. no ABS. The results of this proposed pilot trial will be used to construct a subsequent pivotal prospective, randomized, multi-center clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* This study will recruit adult patients undergoing total hip arthroplasty, lumbar fusion with instrumentation, or femoral-popliteal bypass graft surgical procedures.

Exclusion Criteria:

* The presence of any of the following factors will exclude patients from enrollment in the study:

  1. History of prior prosthesis infection
  2. Active infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2012-01; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rabih O Darouiche, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Michael E. DeBakey VA Medical Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided
Not determined at this time.

REFERENCES:
- [Derived] Darouiche RO, Green DM, Harrington MA, Ehni BL, Kougias P, Bechara CF, O'Connor DP. Association of Airborne Microorganisms in the Operating Room With Implant Infections: A Randomized Controlled Trial. Infect Control Hosp Epidemiol. 2017 Jan;38(1):3-10. doi: 10.1017/ice.2016.240. Epub 2016 Oct 26. PMID 27780479

RESULTS

PARTICIPANT FLOW:
Groups:
- Air Barrier System: The Air Barrier System will be employed throughout the surgical procedure for this group of patients.
  Air Barrier System (Nimbic): ABS is a device that emits a stream of purified air over the surgical site creating a barrier that prevents the intrusion of bacteria.
Period: Overall Study
Arm/Group | Air Barrier System | Control
Started | 150 | 150
Completed | 148 | 146
Not Completed | 2 | 4
Not completed — Surgery not complete | 0 | 1
Not completed — Prosthesis not implanted | 2 | 3

BASELINE CHARACTERISTICS:
Population: A sample size of 150 per group provided a power of 80% to detect a statistically significant 3% difference (alpha<0.05) in surgical site infection rate.
Groups:
- Control: The Air Barrier System will NOT be employed throughout the surgical procedure for this group of patients.
- Total: Total of all reporting groups
Arm/Group | Control | Air Barrier System | Total
Number analyzed (Participants) | 146 | 148 | 294
Age, Customized [Mean (Standard Deviation); unit: years]
  Age in Years | 61.3 (10.4) | 61.1 (9.6) | 61.2 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 138 | 140 | 278
Region of Enrollment [Number; unit: participants]
  United States | 146 | 148 | 294
BMI (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 29.4 (4.5) | 28.8 (5.3) | 29.1 (4.9)
American Society of Anesthesiologists (ASA) Risk Score [Count of Participants; unit: Participants] — The American Society of Anesthesiologists (ASA) risk score is graded on a scale of 1 to 5 (integer), with ASA score of 1 being the least health risk and ASA score of 5 being the greatest health risk.
  ASA score 1: Normal, healthy patient; ASA score 2: Patient with mild, systemic disease; ASA score 3: Patient with severe systemic disease; ASA score 4: Patient with severe systemic disease that is a constant threat to life.
  Participants
    ASA Score 1 | 2 | 0 | 2
    ASA Score 2 | 35 | 39 | 74
    ASA Score 3 | 104 | 105 | 209
    ASA Score 4 | 5 | 4 | 9
History of cardiopulmonary condition [Number; unit: participants]
  Yes | 134 | 139 | 273
  No | 12 | 9 | 21
History of neurological condition [Number; unit: participants]
  Yes | 83 | 85 | 168
  No | 63 | 63 | 126
History of Cancer [Number; unit: participants]
  Yes | 18 | 21 | 39
  No | 128 | 127 | 255
History of diabetes mellitus (type I or II) [Number; unit: participants]
  Yes | 25 | 28 | 53
  No | 121 | 120 | 241
History of smoking [Number; unit: participants]
  Yes | 87 | 109 | 196
  No | 59 | 39 | 98
Number of people in operating room [Mean (Standard Deviation); unit: People in operating room] — Number of people present in operating room at the beginning of each ten-minute interval.
  People in operating room | 8.6 (1.9) | 8.6 (1.8) | 8.6 (1.8)
Surgery time (minutes) [Mean (Standard Deviation); unit: Minutes] | 114.2 (55.0) | 115.8 (60.5) | 115.0 (57.8)
Revision surgery [Number; unit: participants]
  Yes | 13 | 15 | 28
  No | 133 | 133 | 266
Surgery type [Number; unit: participants]
  Total Hip Arthroplasty | 73 | 73 | 146
  Spine Surgery | 66 | 66 | 132
  Vascular Surgery | 7 | 9 | 16
Received preoperative antibiotic prophylaxis [Number; unit: participants]
  Yes | 146 | 148 | 294
  No | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Implant Infection (Number of Occurrences in Each Arm).
Description: Fewer patients in the Air Barrier System group will have implant infection compared to the Control group. Diagnosis of SSI was made by a physician who was masked to the patients' group assignment and not involved in the patients' care by evaluating medical records using the standard and extremely widely used (clinically, epidemiologically, and in research) CDC criteria*, which categorize SSI into superficial incisional, deep incisional, and organ/space/implant levels. Superficial and deep incisional infections were defined and reported as "incisional" infections, whereas organ/space/implant level infections were defined and reported as "implant" infections.
  *See Mangram AJ, et al. Guideline for prevention of surgical site infection, 1999: Hospital Infection Control Practices Advisory Committee. Infect Control Hosp Epidemiol 1999;20:250-278.
Time Frame: One year after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Air Barrier System
Number analyzed (Participants) | 146 | 148
Participants | 4 | 0
Statistical Analysis 1: Comparison: Control vs Air Barrier System; A sample size of 150 per group provided a power of 80% to detect a statistically significant (α≤0.05) 3% difference in SSI rate based on a historical infection rate of 6% in the facility where operations were performed; Test type: Superiority — ABS was expected to be superior to Control; p = 0.067, Regression, Logistic — a priori threshold was 0.05; penalized maximum likelihood (Firth) logistic regression, because infection rate was very low (<3%), as expected; Odds Ratio (OR) = 0.11, 95% CI 2-sided [0.01 to 2.05], Standard Error of Mean 0.16 — The dispersion is the SE of the OR. ABS was the numerator group, Control was the denominator

2. Primary Outcome: Comparison of Levels of Airborne CFU Measured at Incision Sites Between the Control and Air Barrier System Groups
Description: Airborne CFU samplers will be used to monitor bacterial populations at the location immediately adjacent to the surgical site. Air will be drawn through a length of PVC tubing onto agar plates at ten minute intervals. Plates will be incubated for 36 hours at 35 degrees Celsius. Staining and morphological identification will be used to identify and count viable bacteria.
Time Frame: One year post surgery
Measure: Mean (Standard Deviation); unit: CFU/m^3
Arm/Group | Control | Air Barrier System
Number analyzed (Participants) | 146 | 148
CFU/m^3 | 5.3 (7.1) | 2.5 (4.6)

3. Primary Outcome: Percent of Patients With Implant Surgical Site Infection
Description: Patient will be clinically evaluated to identify potential implant SSI through daily visits during the hospital stay, at subsequent clinic visits and hospital stays, or telephonically on a monthly basis for one year. If encounter indicates the potential presence of SSI, physician will make diagnosis of SSI using the CDC criteria. Organ/space/implant level infections were defined and reported as "implant" infections.
Time Frame: Within One Year of Surgical Procedure
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Control | Air Barrier System
Number analyzed (Participants) | 146 | 148
percentage of participants | 2.7 [0.7 to 7.0] | 0 [0 to 2.5]

4. Primary Outcome: Percent of Patients With Incisional Surgical Site Infection
Description: Patient will be clinically evaluated to identify potential incisional SSI through daily visits during the hospital stay, at subsequent clinic visits and hospital stays, or telephonically on a monthly basis for one year. If encounter indicates the potential presence of SSI, physician will make diagnosis of SSI using the CDC criteria. Superficial and deep incisional infections were defined and reported as "incisional" infections.
Time Frame: Within One Year of Surgical Procedure
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Control | Air Barrier System
Number analyzed (Participants) | 146 | 148
percentage of participants | 2.0 [0.4 to 6.0] | 2.7 [0.7 to 6.9]

ADVERSE EVENTS:
Time Frame: One year follow up
Arm/Group | Control | Air Barrier System
Serious Adverse Events (participants affected / at risk) | 0/146 | 0/148
Other Adverse Events (participants affected / at risk) | 0/146 | 0/148

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No